CLINICAL TRIAL: NCT02449486
Title: Ropivacaine Infusion to Alleviate Postoperative Pain After Cardiac Surgery
Brief Title: Ropivacaine After Sternotomy
Acronym: NAROSYD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5070221
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Pain
Keywords: Requirement of postoperative pain medication
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Active Comparator): Ropivacaine 4 ml/h (8 mg/h) continuous infusion for 48 hours
  Interventions: Drug: Ropivacaine
- Placebo (Placebo Comparator): Saline infusion 4 ml/h for 48 hours
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine

SUMMARY:
Continuous ropivacaine infusion to sternotomy wound after coronary artery bypass grafting (CABG) or heart valve surgery to diminish postoperative pain.

DETAILED DESCRIPTION:
A multiporous catheter will be introduced into sternotomy wound to CABG or heart valve surgery patients and continuous ropivacaine infusion 4 ml/h will be started immediately after surgery. Ropivacaine infusion will be administered during 48 postoperative hours. All patients receive patient controlled analgesia (PCA) oxycodone after extubation in the PACU. All patients receive a standardized anesthesia during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG or heart valve surgery patients

Exclusion Criteria:

* Psychic disorders
* Sleep apnea syndrome
* Diabetes mellitus (insulin dependent)
* Obesity, body mass index (BMI) ≥ 35
* Cardiac insufficiency, ejection fraction (EF) ≤ 30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Postoperative oxycodone consumption | 48 postoperative hours
  postoperative PCA administered oxycodone

SECONDARY OUTCOMES:
Pain measured with Visual Analog Scale | 48 postoperative hours
  pain measured with VAS at rest and on movement

CONTACTS AND LOCATIONS:
Overall Officials: Pasi K Lahtinen, MD, PhD, Study Director — Kuopio University Hospital
Locations (1):
- Kuopio University hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No
Data will be published in a peer reviewed medical publication